CLINICAL TRIAL: NCT05788588
Title: A Multi-center, Randomized, Single-blind, Parallel Controlled With Active Drug, Confirmatory Study to Evaluate the Efficacy and Safety of HR19006 Injection for Postoperative Parenteral Nutrition
Brief Title: A Phase Ⅲ Study of HR19006 Injection in Postsurgical Parenteral Nutrition
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HR19006-301
Record Dates: First submitted 2023-03-15; First posted 2023-03-29 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-03

CONDITIONS: Parenteral Nutrition
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Intervention Model Description: Phase Ⅲ, multi-center, randomized, single-blind, parallel controlled with active drug, confirmatory clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HR19006 (Experimental)
  Interventions: Drug: HR19006
- All-in-one parenteral nutrition (Active Comparator)
  Interventions: Drug: All-in-one parenteral nutrition

INTERVENTIONS:
Drug: HR19006 — An emulsion containing the full supply of carbohydrates, amino acids and lipids with a total energy content of 1265kcal in a 1250 ml volume, administered via a central venous line over a time period of approximately 15 hours per day.
  Arms: HR19006
Drug: All-in-one parenteral nutrition — Trial participants are prescribed TPN by the attending physician, which will be administered via a central venous line over a time period of approximately 15 hours per day. The formulation is an emulsion containing the full supply of carbohydrates, amino acids and lipids with a total energy content of 1265kcal in a 1250 ml volume (nitrogen content, heat and liquid quantity as equal as HR19006).
  Arms: All-in-one parenteral nutrition

SUMMARY:
This is a phase Ⅲ, multi-center, randomized, single-blind, parallel controlled with active drug, confirmatory study, and the purpose of the study is to evaluate the efficacy and safety of HR190006 for postoperative parenteral nutrition via central venous catheter.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent;
2. Elective operation of Gastrointestinal;
3. Male or female，aged 18-80 years inclusive;
4. Body Weight at least 40kg, Body mass index (BMI) 18.5-30 kg/m2 inclusive;
5. Nutrition Risk Screening (NRS2002) score at least 3 points.

Exclusion Criteria:

1. Known hypersensitivity to egg-, soy-, and fish proteins or any of the ingredients;
2. Congenital amino acid metabolism abnormality;
3. Hypothyroidism or hyperthyroidism;
4. Significant abnormal values of clinical laboratory examination;
5. Uncompensated hemodynamical failure of any origin (hemorrhagic shock, myocardial infarction, cardiac failure);
6. General contraindications for infusion therapy such as acute pulmonary oedema, hyper-hydration and decompensated cardiac insufficiency;
7. Subjects with a history of mental system diseases and cognitive dysfunction;
8. Serious complications during or after operation;
9. Previous (< 2 weeks) received treatment with intravenous nutrition;
10. Previous (< 4 weeks) or ongoing treatment with growth hormone or corticosteroids;
11. Pregnant or nursing women;
12. No birth control during the specified period of time;
13. Participated in clinical trials of other drugs (received experimental drugs);
14. The investigators determined that other conditions were inappropriate for participation in this clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum prealbumin level on the 6th day after operation. | on day 6 postoperation

SECONDARY OUTCOMES:
The change of serum prealbumin level from baseline on the 6th day after operation. | on days 1 and 6 post operation
The changes of linoleic acid level from baseline on the 6th day after operation. | on days 1 and 6 post operation
The changes of arachidonic acid level from baseline on the 6th day after operation. | on days 1 and 6 post operation
The changes of linolenic acid level from baseline on the 6th day after operation. | on days 1 and 6 post operation
The changes of EPA level from baseline on the 6th day after operation. | on days 1 and 6 post operation
The changes of DHA level from baseline on the 6th day after operation. | on days 1 and 6 post operation
The changes of CRP level from baseline on the 6th day after operation. | on days 1 and 6 post operation
The changes of IL-6 level from baseline on the 6th day after operation. | on days 1 and 6 post operation
The changes of TNF-α level from baseline on the 6th day after operation. | on days 1 and 6 post operation
The incidence of new postoperation infection. | on days 1 and 6 post operation

CONTACTS AND LOCATIONS:
Locations (1):
- Hefei First People's Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided